CLINICAL TRIAL: NCT01423799
Title: Immunonutrition to Improve Quality of Life of Upper Gastrointestinal Cancer Patients Undergoing Oncological Treatment
Brief Title: Immunonutrition and Quality of Life of Cancer Patients Undergoing Oncological Treatment
Acronym: Neoimmune
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 09.54.CLI
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Gastrointestinal Cancer
Keywords: Quality of life; Cancer; Immunonutrition
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasms | interventions — Nucleotides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional product (Experimental): Nutritional intervention containing immuno-nutrients
  Interventions: Dietary Supplement: Nutritional supplements containing arginine, n-3 and nucleotides
- Control Group (Active Comparator): Isocaloric and isonitrogenous control without immuno nutrients.
  Interventions: Dietary Supplement: Isocaloric control

INTERVENTIONS:
Dietary Supplement: Nutritional supplements containing arginine, n-3 and nucleotides — Nutritional intervention with immuno-nutrients
  Arms: Nutritional product
Dietary Supplement: Isocaloric control — Isocaloric and isonitrogenous control without immuno nutrients
  Arms: Control Group

SUMMARY:
The purpose of this study is to compare the health-related quality of life following dietary supplementation with an immunonutrition formulation vs an isocaloric/isoprotein control diet supplement in patients suffering from upper digestive tract neoplasia undergoing oncological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven GI cancer.
* Age ≥ 18 years.
* Life expectancy more than 3 months.
* Female patients of child-bearing potential must be willing to employ effective contraception during the study period.
* Female patients of child-bearing potential must have a negative serum Beta Human Chorionic Gonadotrophin (βhCG) test at Visit 0.
* The patient is able to communicate effectively with study personnel and is considered reliable, willing, and cooperative in terms of compliance with the protocol requirements.
* The patient voluntarily gives written informed consent to participate in the study.

Exclusion Criteria:

* Severe concomitant clinical conditions other than the previously untreated digestive tract cancer that jeopardise the protocol follow-up.
* The patient is pregnant or is a lactating woman.
* Currently participating or having participated in another interventional clinical trial related to nutritional support during the 30 days prior to the beginning of the study product intake, except if this other interventional trial is testing new drug or surgical intervention. (Note: participation in a prior or concurrent clinical trial not related to nutritional support does not exclude the patient from participation.)
* Other malignancies in the last 5 years (except for successfully treated in situ basocellular skin and in situ cervical uterine tumours).
* Patients with more than 20% weight loss over a 6 months period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QOL), measured with the EORTC QLQ-C30 | QOL will me measured 30 days post-surgery

SECONDARY OUTCOMES:
QOL assessed by the EORTC QLQ-OG 25 | QOL will me measured 30 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Mariette, MD, Principal Investigator — University Hospital Claude Huriez, CHRU-Place de Verdun-59037 Lille, Cedex France
Locations (1):
- Centre Hospitalier Régional Universitaire de Lille, Lille, France